CLINICAL TRIAL: NCT04599608
Title: Prediction of Patient Drug Response Using an Ex Vivo Organ Culture (EVOC) on Fresh Human Tumour Samples From Metastatic Patients
Brief Title: Prediction of Drug Response Using an Ex Vivo Organ Culture (EVOC) on Fresh Human Tumour Samples From Metastatic Patients
Acronym: CURESPONSE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Imperial College London (Other)
Collaborators: Curesponse Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20HH6332
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Advanced Cancer; Metastatic Cancer
Keywords: Ex Vivo Organ Culture; Biopsy; Advanced/Metastatic cancer; Prediction of response to cancer treatment
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to determine how sensitive and specific the Curesponse Ex Vivo Organ Culture (EVOC) model is at predicting a patient's clinical response to a specific cancer therapy.

248 patients from participating UK hospitals will have a biopsy for the development of an Ex-vivo organ culture at the Curesponse Laboratory. Patients will have standard of care anticancer therapy after the biopsy and be followed up for 6 months following their biopsy.

The combined results of the study will show whether the EVOC has potential to be useful for future patients prospectively in determining whether a certain clinical treatment is likely to benefit them.

DETAILED DESCRIPTION:
This is a A Phase II multi-centre prediction study of the Curesponse Ex Vivo Organ Culture (EVOC) model in patients with suspected or confirmed advanced or metastatic malignancy.

Patients with suspected or confirmed, advanced or metastatic malignancy in whom at least 1 site is amenable for biopsy, and who would be planned to receive systemic anti-cancer therapy, where disease response can be measured by conventional imaging methods will be recruited for this study.

Patients will undergo a research biopsy where up to 6 tissue samples will be collected. Patients will also have the option to provide an additional single blood sample for germline genetic testing. Patients will then attend their hospital clinical to receive standard of care anticancer therapy as discussed with their oncologist.

Concurrently to the patients treatment, the tissue samples will be transported to the Curesponse laboratory for the development of the EVOC. The EVOC will be treated with a range of anticancer therapies, including the same treatment that the patient will be receiving in clinic. The model will predict whether the cancer will respond to the therapy. Additionally, providing the patient consents, the tissue will also undergo tumour gene profiling related to the secondary and exploratory endpoints and objectives.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected or confirmed advanced or metastatic cancer
2. Aged > 18 years
3. Life expectancy > 3 months
4. ECOG Performance Status 0-2
5. At least one tumour lesion which is amenable for 16 G biopsy (minimum of 2 cores)
6. Planned to receive standard of care therapy or an experimental treatment as part of a clinical trial following the biopsy
7. Written informed consent and ability to comply with study protocol
8. Measurable disease as per Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1 by CT or MRI

Exclusion Criteria:

1. Pregnant and/or breastfeeding woman
2. Lesion is non accessible
3. Any other severe concurrent disease which in the judgment of the investigator would make the patient inappropriate for entry into this study
4. Known carrier for acquired immune deficiency syndrome (AIDS)
5. Known carrier for hepatitis B or hepatitis C virus indicating acute or chronic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected or confirmed, advanced or metastatic malignancy in whom at least 1 site is amenable for biopsy, and who would be planned to receive systemic anti-cancer therapy, where disease response can be measured by conventional imaging methods.
Sampling Method: Non-Probability Sample
Enrollment: 248 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
The EVOC to demonstrate a sensitivity and specificity of at least 70% for predicting a patients clinical response to a specific anti-cancer therapy | From biopsy to the end of the patient's final imaging response assessment at Follow up 3.
  Comparison of patient's treatment clinical to the EVOC treated with the same therapy.
Assessment of tumour heterogeneity in relation to treatment response using the EVOC model | During the biopsy
  Tumour gene profiling on tissue samples obtained at the biopsy
Assess variability in cell populations within the EVOC before and after treatment. | From pre-treatment of EVOC up to the end of treatment on the EVOC model.
  FACS and other methods of analysis to analyse the changes in cell population of the EVOC.
Evaluation and characterisation of viable and resistant cancer cells in the EVOC following treatment and assessment of their response to other therapeutic agents. | End of treatment on EVOC model.
  Following treatment of EVOC, viable/resistant cancer cells to be extracted and harvested, to be further grown for further treatment response assessments in the laboratory.

SECONDARY OUTCOMES:
Comparison of the clinical utility of the EVOC compared to other predictions of response via additional technologies for cancer treatment. | Biopsy up to end of treatment of EVOC.
  Assessed by genomic profiling where relevant, and the comparison of tumour gene profiling to germline genetic testing.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Krell, Dr, Principal Investigator — Imperial College London